CLINICAL TRIAL: NCT05965024
Title: Exploration on the Value of Molecular Residual Disease Based on Circulating Tumor DNA Detection in Predicting Recurrence of Resected Non-small Cell Lung Cancer
Brief Title: Exploration on the Value of MRD Based on ctDNA Detection in Predicting Recurrence of Resected Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: LungMate-016
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the unique patented MONOD and Methyl Titan methylation sequencing technology on lung cancer tissue and blood samples, a lung cancer MRD monitoring panel is designed. The panel is used to detect molecular residual disease of stage IB-IIIB non-small cell lung cancer patients underwent radical surgery, explore personalized analysis models, and conduct research on recurrence monitoring for non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Patients with pathological diagnosis of non-small cell lung cancer and clinical staging of stage IB-IIIB;
3. Able to undergo radical surgical treatment;
4. Physical condition score (ECOG) ≤1;
5. The expected survival time exceeds 24 months;
6. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Individuals with a history of other malignant tumors within 5 years;
2. Those who have undergone neoadjuvant therapy before surgery;
3. Postoperative incision margin R1 or incision margin R2;
4. Those who have undergone a blood transfusion within 2 weeks before the surgery;
5. Individuals with systemic inflammatory response syndrome;
6. Those with serious diseases of important organs such as the heart, lungs, kidneys, and brain;
7. Participants in other clinical trials within the past 30 days and have taken investigational drugs;
8. Due to various reasons, sampling cannot be completed, samples do not meet the requirements, or baseline samples (preoperative and postoperative plasma samples, tumor tissue samples) are incomplete;
9. Researchers believe that it is not appropriate to participate in this experiment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with pathological diagnosis of non-small cell lung cancer and clinical staging of stage IB-IIIB
Sampling Method: Non-Probability Sample
Enrollment: 377 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | Up to 24 months
  Recurrence-free survival means the time from the date of surgery to the first recorded date of disease recurrence or patient death, whichever occurs earlier. 2-year recurrence-free survival rate means the rate of patients survive without recurrence for 2 years or more.

SECONDARY OUTCOMES:
Median recurrence-free survival | up to 60 months
  Recurrence-free survival means the time from the date of surgery to the first recorded date of disease recurrence or patient death, whichever occurs earlier. Median recurrence-free survival means the median value of recurrence-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided